CLINICAL TRIAL: NCT02679157
Title: Prognostication of Need for Rehabilitation and Special Support in ICU Survivors. Two Studies Prognosticating Adverse Physical or Psychological Outcome
Brief Title: Prognostication of Need for Rehabilitation and Special Support in ICU Survivors
Acronym: PROGRESS-ICU
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Peter Sackey, Associate professor, Karolinska Institutet
Other Study IDs: EPN 2015/1799-31
Record Dates: First submitted 2016-01-28; First posted 2016-02-10 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Physical Disability; Depression; Posttraumatic Stress Disorder; Anxiety
Keywords: Posttraumatic stress disorder; Depression; Anxiety; ADL; Health-related quality of life; ICU survivorship
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Title: PROGnostication of need for REhabilitation and Special Support after Intensive Care Unit Stay - a multinational, observational study

Objectives:

1. To investigate associations between potential risk factors (premorbid factors, in-ICU treatments/diagnoses and patient status at ICU discharge) and three-month physical and psychological outcome in ICU survivors.
2. Based on the associations between identified risk factors and adverse outcomes, create and validate instruments, to be used at ICU discharge, predicting new-onset physical or psychological problems three months after ICU discharge.

Study design:

Prospective, observational multi centre (10 centres) cohort studies

Outcomes:

Adverse psychological outcome three months after ICU discharge (Posttraumatic Stress Syndrome-14 (PTSS-14) part B score >45 or Hospital Anxiety and Depression Scale (HADS) subscale score >10). New-onset physical disability, defined as a reduction in Barthel Index ≥10 points compared with 2 weeks prior to hospital admission.

Study duration:

Recruitment of patients during 2-4 months in the ten study sites. Follow-up of primary endpoints 3 months after ICU discharge.

Number of subjects:

The aim is to screen all eligible patients and include 600-1000 ICU survivors during the recruitment period. The final number of included patients depends on case-mix in the units and potential exclusions.

Population:

Adult patients (18 years or older) discharged from ICU.

DETAILED DESCRIPTION:
Every year, an estimated 5 million patients are treated in European Intensive Care Units (ICUs) yearly, with 40 000 in Swedish ICUs alone (1,2). As many as 50 % of ICU survivors suffer from new-onset physical, psychological or cognitive problems in the months or even years after ICU discharge, irrespective of the reason for ICU admission (3-5). These problems are major hurdles for patients discharged from the ICU to return to life as it was prior to hospitalisation, but often remain unrecognised by healthcare providers (3-5). Follow-up led by ICU clinicians is increasingly recognised as an addendum to critical care (5,6). Yet, interventions in large and unselected groups of ICU survivors have failed to demonstrate meaningful improvements (7,8) except in vulnerable subgroups (9,10). Dilution of treatment effects is a recognised problem in interventional studies (11). Thus, identifying patients with risk for adverse outcome is an important enrichment step prior to evaluation of new interventions. The importance has recently been highlighted at a stakeholders meeting regarding post-ICU syndrome (12). Pilot studies from our research group indicate that risk prediction instruments for ICU survivors with fairly good accuracy can be developed and used in clinical practice (13,14) but predictors need to be assessed and validated in a larger sample.

Data collection All data will be entered in coded form to a web-based, electronic Case Report Form (Pheedit eCRF) supplied by the Central Steering Committee. The eCRF will be accessible with a username and password at all computers with internet access. All data can be entered in the eCRF. Each centre will keep a safely placed and locked patient ID and study code list, separate from the study data.

Potential risk factors:

Patient characteristics Age Sex Educational level** Working/school/parental leave/retired/unemployed/sick-leave** Physical comorbidities (Charlson Comorbidity Index & SAPS III box 1) (supplement) History of psychological problems before ICU stay, including substance abuse) Caretaker of a child <18 years old** Barthel Index-100 prior to falling ill, reported by patient, and/or proxy together with medical chart review

In-ICU diagnoses/treatments/status Admission diagnosis (medical/surgical/trauma) Acute/elective hospital admission Admission severity of illness (APACHE II) Pelvic fracture Fractures (other than pelvic) ICU length of stay (hours) Severe sepsis/septic chock* Days with coma (for any reason) Days with invasive ventilator treatment Agitation/agitated delirium during ICU stay**

Patient status at ICU discharge Depressive symptoms with PHQ2 questions (two questions, supplement)** Chelsea Critical Care Physical Assessment Tool (CPAx) Questions 1-5 (supplement) within 24 hours prior to discharge* PTSS-14 Part A (four questions, supplement)** Social support (one question, supplement)

Three months post-ICU discharge Hospital Anxiety and Depression Scale (HADS) (supplement) Posttraumatic Stress Symptoms 14 (PTSS-14) (supplement) Barthel Index (supplement) Short Form 36 Health Survey (supplement) Health utilization questionnaire

Questionnaires will be sent by postal mail to all patients, together with an information letter about participation in the studies and a consent form to sign for those unable to give consent at inclusion. A phone number will be supplied, for patients with questions or who wish to know more regarding their ICU stay. Ten-fourteen days after questionnaires have been sent out, a reminder telephone call will be made to patients who have not returned the questionnaires.

Consent Patients will be asked for consent at study inclusion. If unable to consent, patients will be asked for consent at three months post ICU, when questionnaires are being sent out.

Inter-rater reliability Risk factors that are assessed by observation, where no validated instruments are available, will undergo interrater reliability testing within the study. Ten patients per centre will be assessed in parallel by two independent observers, blinded to each other´s assessment. Specifically, the factors are the items of CPAx.

Outcome measures:

Two primary outcome measures:

1. Adverse psychological outcome at three months post-ICU discharge is defined as a subscale score >10 in the Hospital Anxiety and Depression Scale (HADS), indicative of clinically significant depressive or anxiety symptoms, AND/OR a Posttraumatic Stress Symptoms -14 (PTSS-14) part B score >45 indicative of clinically significant posttraumatic stress symptoms.
2. Adverse physical outcome (new-onset physical disability) three months post-ICU discharge is defined as a worsening of the Barthel Index-100 by 10 points or more, compared to the reported Barthel Index-100 two weeks prior to hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

ICU stay>24 hours for postoperative patients and >12 hours for other ICU admissions

Exclusion Criteria:

1. Previously documented cognitive impairment (e.g. dementia or intellectual development disorder resulting in poor understanding/compliance in outcome assessment)
2. No home address
3. Unable to read and write in language spoken at local study site (Swedish/Danish/Dutch)/used in questionnaires
4. Patient declines participation
5. Moribund patient or with more than one limitation of therapy
6. Need for neurointensive care due to head trauma, intracranial hemorrhage or infarction AND GCS never better than 13 in the first 48 hours
7. Transfer to other ICU before discharge to ward
8. Solely in ICU for elective procedure (eg central line, epidural)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 573 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Adverse psychological outcome | Three months post-ICU
  Caseness defined as PTSS-14 part B score above 45 or HADS subscale score above 10
Adverse physical outcome | Three months post-ICU
  Caseness defined as Reduction in Barthel Index (0-100) by 10 points or more

SECONDARY OUTCOMES:
Health-related quality of life assessed with Short Form -36 in patients | In first three months post-ICU
  Health-related quality of Life domains in relation to adverse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Sackey, MD, PhD, Study Chair — Karolinska University Hospital; Anna Milton, MD, Principal Investigator — Karolinska University Hospital
Locations (10):
- Denmark (2):
  - Rigshospitalet Copenhagen, Copenhagen
  - Odense University Hospital, Odense
- Netherlands (2):
  - University Medical Centre Radboud, Nijmegen
  - University Medical Centre Utrecht, Utrecht
- Sweden (6):
  - Östersund Hospital, Östersund, Jämtland County
  - Umeå University Hospital, Umeå, Västerbotten County
  - Örebro University Hospital, Örebro
  - Dept of Anesthesiology, Surgical Services and Intensive Care Medicine, Karolinska University Hospital, Stockholm
  - Stockholm South Hospital, Stockholm
  - Dept of Anesthesia and Intensive Care, Uppsala Akademiska, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhodes A, Ferdinande P, Flaatten H, Guidet B, Metnitz PG, Moreno RP. The variability of critical care bed numbers in Europe. Intensive Care Med. 2012 Oct;38(10):1647-53. doi: 10.1007/s00134-012-2627-8. Epub 2012 Jul 10. PMID 22777516
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Desai SV, Law TJ, Needham DM. Long-term complications of critical care. Crit Care Med. 2011 Feb;39(2):371-9. doi: 10.1097/CCM.0b013e3181fd66e5. PMID 20959786
- [Background] Modrykamien AM. The ICU follow-up clinic: a new paradigm for intensivists. Respir Care. 2012 May;57(5):764-72. doi: 10.4187/respcare.01461. Epub 2011 Dec 8. PMID 22152275
- [Background] Cuthbertson BH, Rattray J, Campbell MK, Gager M, Roughton S, Smith A, Hull A, Breeman S, Norrie J, Jenkinson D, Hernandez R, Johnston M, Wilson E, Waldmann C; PRaCTICaL study group. The PRaCTICaL study of nurse led, intensive care follow-up programmes for improving long term outcomes from critical illness: a pragmatic randomised controlled trial. BMJ. 2009 Oct 16;339:b3723. doi: 10.1136/bmj.b3723. PMID 19837741
- [Background] Jones C, Skirrow P, Griffiths RD, Humphris GH, Ingleby S, Eddleston J, Waldmann C, Gager M. Rehabilitation after critical illness: a randomized, controlled trial. Crit Care Med. 2003 Oct;31(10):2456-61. doi: 10.1097/01.CCM.0000089938.56725.33. PMID 14530751
- [Background] Schandl A, Bottai M, Hellgren E, Sundin O, Sackey P. Gender differences in psychological morbidity and treatment in intensive care survivors--a cohort study. Crit Care. 2012 May 14;16(3):R80. doi: 10.1186/cc11338. PMID 22578016
- [Background] Schandl A, Bottai M, Hellgren E, Sundin O, Sackey PV. Developing an early screening instrument for predicting psychological morbidity after critical illness. Crit Care. 2013 Sep 24;17(5):R210. doi: 10.1186/cc13018. PMID 24063256
- [Background] Schandl A, Bottai M, Holdar U, Hellgren E, Sackey P. Early prediction of new-onset physical disability after intensive care unit stay: a preliminary instrument. Crit Care. 2014 Jul 31;18(4):455. doi: 10.1186/s13054-014-0455-7. PMID 25079385
- [Background] Sackett DL. Why randomized controlled trials fail but needn't: 2. Failure to employ physiological statistics, or the only formula a clinician-trialist is ever likely to need (or understand!). CMAJ. 2001 Oct 30;165(9):1226-37. No abstract available. PMID 11706914
- [Derived] Milton A, Schandl A, Soliman IW, Meijers K, van den Boogaard M, Larsson IM, Brorsson C, Ostberg U, Oxenboll-Collet M, Savilampi J, Paskins S, Bottai M, Sackey PV. Development of an ICU discharge instrument predicting psychological morbidity: a multinational study. Intensive Care Med. 2018 Dec;44(12):2038-2047. doi: 10.1007/s00134-018-5467-3. Epub 2018 Nov 22. PMID 30467678
- See also: NICE Guidelines for ICU follow-up — http://www.nice.org.uk/CG83